CLINICAL TRIAL: NCT02493218
Title: D-Stress Baltimore: School-based Mindfulness Instruction for Primary Prevention of Mental Health and Behavioral Problems in Middle School
Brief Title: D-Stress Baltimore: School-based Mindfulness Instruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Elev8 Baltimore (Other); Abell Foundation (Other); University of Chicago (Other); Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: NA_00077391
Record Dates: First submitted 2015-06-26; First posted 2015-07-09 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Coping; Stress Disorders, Post-Traumatic; Mental Health Wellness 1
Keywords: mindfulness; intervention; african american; youth; stress; poverty
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness Instruction (Experimental): Instruction on mindfulness concepts and practices. Classes are 45-90 minutes each and held weekly for 12 weeks.
  Interventions: Behavioral: Mindfulness Instruction
- Health Education Instruction (Active Comparator): Instruction on general health and wellness. Classes are 45-90 minutes each and held weekly for 12 weeks.
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Mindfulness Instruction — Age-appropriate instruction on mindfulness concepts and practices, adapted from the mindfulness-based stress reduction (MBSR) program. Classes are 45-90 minutes each and held weekly for 12 weeks.
  Arms: Mindfulness Instruction
Behavioral: Health Education — Age-appropriate health education concepts and topics. Classes are 45-90 minutes each and held weekly for 12 weeks.
  Arms: Health Education Instruction

SUMMARY:
Effective strategies to ameliorate the negative effects of stressful urban living are greatly needed. D-Stress Baltimore (DSB) is an evidence-based mindfulness-based instructional program of stress-reduction techniques, found to reduce mental health problems across many adult populations.

The investigators propose to conduct a randomized controlled trial of the 12-week school-based DSB program compared with a 12-week school-based health education control program at Elev8 schools among 5th-8th graders to assess if DSB program is beneficial for mental health and behavioral problems among public middle-school students.

DETAILED DESCRIPTION:
Urban youth in Baltimore City are under significant and inevitable stresses, including violent neighborhoods, failing schools, and interpersonal conflict. Effective strategies to ameliorate the negative effects of stressful urban living are greatly needed.

D-Stress Baltimore (DSB) is an evidence-based mindfulness-based instructional program of stress-reduction techniques which has been found to be beneficial for adults in decreasing anxiety and depression, improving positive emotions, and reducing anger.

The investigators propose to conduct a randomized controlled trial of the 12-week school-based DSB program compared with a 12-week school-based health education control program at Elev8 schools among 5th-8th graders. The investigators hypothesize that the D-Stress Baltimore Program will reduce negative emotions, including hostility, and improve coping.

ELIGIBILITY:
Inclusion Criteria:

* 5th - 8th graders in select Baltimore City schools

Exclusion Criteria:

* N/A

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 400 (Actual)
Dates: Start 2012-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | 9 months
  Assessment of impact of Mindfulness instruction versus Health Education instruction as measured by scores on mental health questionnaire administered at baseline, and then 3 and 9 months later. Children's Depression Inventory - Short Form (CDI-S)
Affect Measures: Positive and Negative Affect Scale; State Trait Anger Expressivity Index; Differential Emotions Scale | 9 months
  Assessment of impact of Mindfulness instruction versus Health Education instruction as measured by scores on mental health questionnaire administered at baseline, and then 3 and 9 months later.
Anxiety assessed by Multidimensional Anxiety Scale of Childhood. | 9 months
  Assessment of impact of Mindfulness instruction versus Health Education instruction as measured by scores on mental health questionnaire administered at baseline, and then 3 and 9 months later.

SECONDARY OUTCOMES:
Coping Questionnaire | 9 months
  Assessment of impact of Mindfulness instruction versus Health Education instruction on coping as measured by scores on questionnaire administered at baseline, and then 3 and 9 months later. Specific coping measures used are: Brief COPE Inventory; the Coping Self-Efficacy Scale (CSE); and Children's Response Style Questionnaire (CRSQ).
Post-traumatic stress symptoms | 9 months
  Assessment of impact of Mindfulness instruction versus Health Education instruction as measured by scores on questionnaire administered at baseline, and then 3 and 9 months later.
  Children's Post-traumatic Stress Symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Erica Sibinga, MD, MHS, Principal Investigator — Johns Hopkins School of Medicine
Locations (3):
- United States (3):
  - Tench Tilghman Elementary Middle School, Baltimore, Maryland
  - Collington Square Elementary Middle School, Baltimore, Maryland
  - Commodore John Rodgers Elementary Middle School, Baltimore, Maryland

REFERENCES:
- [Derived] Sibinga EM, Webb L, Ghazarian SR, Ellen JM. School-Based Mindfulness Instruction: An RCT. Pediatrics. 2016 Jan;137(1). doi: 10.1542/peds.2015-2532. Epub 2015 Dec 18. PMID 26684478